CLINICAL TRIAL: NCT06419972
Title: Effectiveness of a Combined Education and Exercise Program on the Physical, Functional and Psychological Status of Climacteric Women.
Brief Title: Multimodal Program for Climacteric Women
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Valencia (Other)
Responsible Party: Principal Investigator, Laura Fuentes Aparicio, Assistant Professor of Physiotherapy, University of Valencia
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: UV_Menopause
Record Dates: First submitted 2024-05-07; First posted 2024-05-17 (Actual); Last update posted 2025-02-03 (Actual); Status verified 2025-01

CONDITIONS: Climacteric Syndrome; Postmenopausal Symptoms; Menopause; Perimenopausal Disorder
Keywords: perimenopause; climacteric; Postmenopause; women's health

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): They will receive multimodal physiotherapy programme, which will combine therapeutic exercise based in general strength exercise combined with a pelvic floor education program.
  Interventions: Other: multimodal physiotherapy programme
- Control (No Intervention): They will not receive any type of intervention

INTERVENTIONS:
Other: multimodal physiotherapy programme — The intervention to which the climacteric women will be subjected will consist of a combined program of education and general strength and pelvic floor muscles exercises of 8 weeks duration, at a rate of 2 sessions/week. Each of the sessions will last 60 min, except for the first one, which will be 90 min.
  Arms: Experimental

SUMMARY:
Your study seems to aim at emphasizing the significance of non-pharmacological and non-hormonal approaches in managing menopausal symptoms, particularly focusing on muscle training and education. This holistic approach acknowledges the importance of physical well-being, psychological support, and education to enhance women's quality of life during the menopausal transition.

DETAILED DESCRIPTION:
Climacteric is a time of great transition for all women physically, mentally, and emotionally . This transition involves a host of physical, endocrine, and psychological changes that are influenced by ethnic, psychological, and sociocultural factors . Each woman's experience of the menopausal transition is unique; therefore, a one-size-fits-all approach to symptom management is not sufficient .

Menopause is a retrospective diagnosis and is said to occur when menstrual activity has ceased for at least 12 consecutive months with no other physiologic or pathologic explanation for it . It marks the end of reproductive life and ovarian follicular activity by the onset of an estrogen deficiency that triggers various symptoms .

The main symptoms aggregated according to the Menopause Rating Score MRS include somatic symptoms [vasomotor symptoms (hot flashes and night sweats), sleeping difficulties, fatigue, palpitations, joint pain, worsening muscle ability and function, skin/eye dryness, and skin and hair changes], psychological [mental confusion, mood swings, increased anxiety, irritability], and urogenital [genitourinary syndrome symptoms (vaginal dryness, dyspareunia, irritation, itching, sexual dysfunction), bladder symptoms (altered frequency, level of urgency and incontinence).

Focusing on the musculature and ligaments, we must also think about the tissues of the pelvic floor muscle (PFM), which are affected by the drop in estrogen levels, due to the existence of estrogen receptors in ligaments, musculature and pelvic support structures. The pelvic floor as a whole has an important role in supporting the organs of the pelvic cavity and is involved in the closing and opening mechanisms of the urethral, vaginal and anal tract . Taking this into account, what can be worked on voluntarily is the musculature.

This estrogenic variation is also responsible for the onset of cardiovascular disease during the menopausal period, which is characterized by variations in the lipid profile and the predominant accumulation of abdominal fat.

Treatments to treat menopausal symptoms include hormonal preparations, non-hormonal medications and non-pharmacological therapies. The latter two, non-pharmacological and non-hormonal therapies are generally the least studied.

On genitourinary and urinary syndrome symptoms, the musculature has a fundamental role, and working on it will produce improvements in these factors. By training the pelvic floor muscle (PFM) there is a greater blood supply, which this will lead to a relaxation of the tissues and an increase in elasticity that will help in the genitourinary syndrome; and on the other hand, its training, increasing strength, will improve the control and efficacy of the closing and opening of the urethral, vaginal and anal tracts .

On the other hand, physical activity will help in weight loss and improve body composition parameters .

It should be noted that the information provided to women influences the understanding and how menopause and its symptoms are faced, being relevant to provide knowledge and education by the general practitioner or a qualified health personnel.

Therefore, this study seeks to expand the information on non-pharmacological and non-hormonal therapies, such as active training of the pelvic floor muscle, generic muscle training and education, due to their potential efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Women aged ≥45 years
* Women in climacteric period

Exclusion Criteria:

* Musculoskeletal, cognitive, infectious, neurological, or cardiorespiratory pathology impairing assessment or program completion.
* Surgical intervention in lumbopelvic or gynecological region within the last 6 months.

Undergoing oncological treatment.

* Also included women with stable hormone replacement therapy for at least the last 6 months.

Ages: 45 Years to 85 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 115 (Estimated)
Dates: Start 2024-05-30 (Actual); Primary Completion 2025-03-25 (Estimated); Study Completion 2025-06-28 (Estimated)

PRIMARY OUTCOMES:
Upper limb muscle strength | 8 weeks (2 assessment times: T1(pre-intervention), T2 (Immediately post-intervention)and T3 (3-months follow-up)
  For performed the upper limb muscle strength (kg) evaluation will use different dynamometry test
  Dynamometry of Upper limb muscle: using the Hand grip strength (stable position - elbow 90º and arm in contact with the trunk , hold dynamometer with the hand and perform maximum grip force for 5seconds.
Lower limb muscle strength | 8 weeks (2 assessment times: T1(pre-intervention), T2 (Immediately post-intervention)and T3 (3-months follow-up)
  The quadriceps dynamometry test (Lafayette Instrument) will be used to evaluate the muscular strength of the lower extremities, the unit of measure will be. The Lafayette measuring range is 0-300 lbs (136.1 kg/1335 N).
Trunk flexor isometric strength | 8 weeks (2 assessment times: T1(pre-intervention), T2 (Immediately post-intervention)and T3 (3-months follow-up)
  For the isometric strength of the trunk flexors, the central dynamometry test (Lafayette Instrument) will be used: the patient will be in the supine position with the knees straight, the hips flexed at 30° and the trunk at 30°; placing the dynamometer on the sternum, below the suprasternal notch, the participants should place their hands on the opposite acromion processes.The Lafayette measuring range is 0-300 lbs (136.1 kg/1335 N).
Abdominopelvic muscle function | 8 weeks (2 assesment times: T1(pre-intervention), T2 (Immediately post-intervention)and T3 (3-months follow-up)
  The Supine Bridge Test involves lying on a mat with knees and hips flexed, lifting the pelvis off the floor for alignment. The Prone Bridge requires lying face down on elbows, lifting the pelvis so only forearms and toes touch the floor. In the Side Bridge, one lies on their side, supporting the body with elbow, forearm, and feet while lifting the hips. Participants hold each position as long as possible to assess core strength and stability.
Abdominal ultrasound image | 8 weeks (2 assesment times: T1(pre-intervention), T2 (Immediately post-intervention) and T3 (3-months follow-up)
  Will be measure abdominal wall thickness at rest and during a draw-in maneuver for Transversus abdominis (TrA), obliquus internus (IO), and obliquus externus (EO) on the dominant side. Subjects will lie supine with hips and knees flexed. Using a 5.3-10 MegaHertz (MHz) linear probe, the transducer will be centered transversely just above the iliac crest at the umbilical level and aligned with the axillary midline. Three measurements will be taken at each point, averaged for analysis, with the M-line set to the midline for precise measurements. Changes in muscle thickness (cm) reflecting muscle activation will be observed.
Pelvic floor muscle ultrasound image | 8 weeks (2 assesment times: T1(pre-intervention), T2 (Immediately post-intervention) and T3 (3-months follow-up)
  Transabdominal ultrasound will be used, for this purpose convex probe will be place at suprapubic level in B-mode will be used (3.5-5MegaHertz (Mhz). Three measurements at each point and use the mean of the 3 for subsequent analyses. Changes in muscle thickness refected by muscle activation will be calculated as the thickness during contraction minus the resting thickness (cm) .
30s chair-stand test | 8 weeks (2 assesment times: T1(pre-intervention), T2 (Inmediately post-intervention) and T3 (3-months follow-up)
  Women will start from a seated position with feet flat on the floor and arms crossed, rise completely with hips and knees extended, then sit back down touching the seat, repeat for 30 seconds. Chair leaning against a wall, usual footwear. If unable to stand, hands can be placed on legs or mobility aids can be used, scored as adapted test. It is recommended to practice 2-3 slow repetitions for comprehension. Scoring: Count the total number of complete bipedestation (up and down) in a test. If at least one bipedestation is completed in 30 seconds, it is counted. If unable to stand, the score is zero. Record the adapted score if applicable.
Pelvic floor muscles strength | 8 weeks (2 assesment times: T1(pre-intervention), T2 (Immediately post-intervention)
  Vaginal palpation will be done using the Modified Oxford Scale, which comprises 6 levels. It demonstrates good interobserver reliability and serves as a subjective scale for clinical rather than research purposes. To gauge sensitivity to change, each point was supplemented with a +/-, expanding the scale to include 15 degrees.
Pelvic floor muscles Dynamometry | 8 weeks (2 assesment times: T1(pre-intervention), T2 (Immediately post-intervention) and T3 (3-months follow-up)
  A commercially available instrumented plastic dynamometric speculum (Pelvimeter, Phenix, Montpellier, France) was utilized to measure pelvic floor muscle (PFM) tone and maximum intravaginal pelvic floor muscle (PFM) strength generated through maximal voluntary contraction the measure will be reported in grams. All numerical values of pelvic floor muscle (PFM) dynamometry tone are presented as raw values, including the ambient pressure value (170 g). Latex or polyethylene protective covers were used, and the dynamometer was comfortably aligned in the participant's vaginal canal throughout the experiment. Pelvic floor muscle strength was calculated as the mean of three maximum voluntary contractions.

SECONDARY OUTCOMES:
Menopause symptoms | 8 weeks (2 assesment times: T1(pre-intervention), T2 (Immediately post-intervention) and T3 (3-months follow-up)
  The Menopause Rating Scale (MRS) is a widely used tool for assessing symptoms related to menopause.
  The scoring scheme increases point by point with increasing subjectively perceived symptom severity for each of the 11 items (severity 0 [no complaint] to 4 score points [very severe symptoms]). The composite score for each of the dimensions (subscales) is based on the sum of the scores for each item of the respective dimensions. The composite score (total score) is the sum of the dimension scores.
Psychologic condition | 8 weeks (2 assessent times: T1(pre-intervention), T2 (Immediately post-intervention) and T3 (3-months follow-up)
  The Beck Depression Inventory (BDI) is a widely used self-report inventory for measuring the severity of depression symptoms. It consists of 21 multiple-choice questions, each assessing a different symptom of depression such as sadness, pessimism, guilt, and suicidal thoughts. Respondents rate the severity of each symptom over the past two weeks. Scores are summed to yield a total score, with higher scores indicating more severe depressive symptoms. The BDI is frequently used in clinical and research settings to assess depression severity and monitor treatment progress.
Urinary symptoms | 8 weeks (2 assesment times: T1(pre-intervention), T2 (Immediately post-intervention)
  The Pelvic Floor Distress Inventory-20 (PFDI-20) is a recommended questionnaire for evaluating pelvic floor disorder (PFD) symptoms and measuring their impact on women's quality of life. This questionnaire is validated in Spanish. The PFDI-20 reflects different perspectives, thus including 20 questions divided into three symptom scales: pelvic organ prolapse symptoms (POP-DI) (questions 1 to 6); colorectal-anal symptoms (CRADI) (questions 7-14); and urinary symptoms (UDI) (questions 15-20). The questions in the CRADI scale are about fecal incontinence (FI), except for question 11, which addresses flatulence incontinence; whereas the UDI scale addresses urinary symptoms specifically. Question 16 pertains to urgency urinary incontinence (UUI), and question 17 pertains to stress urinary incontinence (SUI). Each question can be answered on four levels of dysfunction: none, mild, moderate, and severe.
Pelvic floor health knowledge | 8 weeks (2 assesment times: T1(pre-intervention), T2 (Immediately post-intervention) and T3 (3-months follow-up)
  Pelvic Floor Impact Questionnaire (PIKQ)It is a tool used to assess the impact of pelvic floor disorders, such as urinary incontinence, colorectal-anal symptoms, and genital prolapse, on various aspects of a person's life, including activities, relationships, and emotions. The questionnaire consists of seven questions for each symptom category (urine, colorectal-anal, and genital prolapse), with responses rated on a scale of none, mild, moderate, or severe. The total score is calculated by summing the scores from each category, with a maximum possible score of 300.

CONTACTS AND LOCATIONS:
Locations (2):
- Spain (2):
  - Department of Physiotherapy. University of Valencia, Valencia
  - Laura Fuentes Aparicio, Valencia

IPD SHARING:
Plan to Share IPD: No